CLINICAL TRIAL: NCT05805098
Title: Venetoclax in Combination With Homoharringtonine and Cytarabine in Newly Diagnosed Subjects With Acute Myeloid Leukemia: a Phase 2/3, the Single-arm, Open-label, Monocentric Study
Brief Title: Venetoclax Combined With Homoharringtonine and Cytarabine in Induction for AML
Acronym: VHA
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SZQ001
Record Dates: First submitted 2023-03-28; First posted 2023-04-07 (Actual); Last update posted 2023-04-07 (Actual); Status verified 2023-03

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — venetoclax; Homoharringtonine; Cytarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Venetoclax Combined With Homoharringtonine and Cytarabine (Experimental): All recipients in this arm received Venetoclax, Homoharringtonine and Cytarabine. Venetoclax was uesd as 100 mg on day 1, 200 mg on day 2, 400mg from day-3 to day-28. Homoharringtonine was uesd as 1 mg/m2 qd from day-1 to day-5. Cytarabine was uesd as 100 mg/m2 qd from day-1 to day-5.
  Interventions: Drug: Venetoclax; Drug: Homoharringtonine; Drug: Cytarabine

INTERVENTIONS:
Drug: Venetoclax — Starting on day 1, venetoclax will be dose escalated to a target dose of 600 mg in the following manner: 100 mg on day 1, 200 mg on day 2 and 400 mg on day 3. The patient then continues to take the 400mg dose for the remainder of the 28 day cycle. Each dose of venetoclax will be self-administered with approximately 240 mL of water within 30 minutes after the completion of a meal, preferably breakfast. The dose should be administered at the same time each day.
  Other Names: VEN
Drug: Homoharringtonine — On day 1, homoharringtonine 1 mg/m2 IV will be given, and will continue for 5 days.
  Other Names: HHT
Drug: Cytarabine — On day 1, cytarabine 100 mg/m2 IV will be given, and will continue for 5 days.

SUMMARY:
This study aims to evaluate the efficacy and safety of venetoclax combined with homoharringtonine and cytarabine in the treatment of newly diagnosed acute myeloid leukemia.

DETAILED DESCRIPTION:
This is a phase II/III study that seeks to treat patients ages 18-60 who have acute myeloid leukemia but have never been treated before. In order to improve the outcome of patients with primary AML, venetoclax combined with homoharringtonine and cytarabine was applied in the treatment of primary AML. This study aims to evaluate the efficacy and safety of venetoclax in combination with homoharringtonine and cytarabine in newly diagnosed subjects with AML.Depending on the level of recovery, patients will either be forced to come off study or have the option to continue the medication, receive maintenance therapy, or pursue an allogeneic stem cell transplant. After completion of study treatment, participants are followed up every 3 to 6 months for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who sign the informed consent must have the ability to understand and be willing to participate in the study and sign the informed consent.
2. patients must have confirmation of AML by WHO criteria, previously untreated, and eligible for treatment with intensive chemotherapy as defined by the following: Cardiac history of congestive heart failure requiring treatment or ejection fraction ≤ 50% or chronic stable angina. Diffusing capacity of the lung for carbon monoxide (DLCO) ≤ 65% or forced expiratory volume during the first second (FEV1) ≤ 65%. Creatinine clearance < 45 mL/min. Moderate hepatic impairment with total bilirubin > 1.5 × ULN. Any other comorbidity that the physician judges to be incompatible with intensive chemotherapy.
3. Patients > 18 to ≤ 60 years
4. Eastern Cooperative Oncology Group (ECOG) Performance Status of ≤2
5. Laboratory values meeting the following criteria:Creatinine clearance ≥ 45 mL/min calculated by the Cockcroft Gault formula or measured by 24-hour urine collection, Serum aspartate aminotransferase (AST) ≤ 3.0 × upper limit of normal (ULN) 、Serum alanine aminotransferase (ALT) ≤ 3.0 × ULN (Unless considered due to leukemic organ involvement), Total bilirubin ≤ 1.5 × ULN, White blood cell (WBC) count < 25 × 109 /L (hydroxyurea is permitted to meet this criterion)

Exclusion Criteria:

1. > 60 years of age or <18 years of age
2. Acute promyelocytic leukemia (M3)
3. Patient is ineligible for treatment with intensive chemotherapy
4. Patient with active infection not controlled, active bleeding from vital organs
5. Patient with history of clinically significant drug or alcohol abuse that would adversely affect evaluation in this study
6. Patient has any other significant medical or psychiatric history that in the opinion of the investigator would adversely affect participation in this study.
7. Female who are pregnant, breast feeding or childbearing potential without a negative urine pregnancy test at screen.
8. Patients with uncontrolled infection with human immunodeficiency virus (HIV) or active Hepatitis B or C
9. Patients deemed unsuitable for enrolment by the investigator.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2028-03-01 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (ORR) | 28 days after study treatment
  Defined as complete response (CR) + CR with incomplete blood count recovery (CRi) + morphologic leukemia-free state (MLFS) + partial response (PR).

SECONDARY OUTCOMES:
Rate of Participants With Adverse Events | Through 28 days post study medication administration
  Percentage of Participants with 3 or 4 grade Adverse Events reported through 28 days post study medication administration.
Event-free survival | Through study completion, up to 3 years
  Defined as the number of days from the date of treatment initiation (i.e., course 1 day 1) to the date of documented treatment failure, relapses from CR, or death from any cause, whichever occurs first. Will be calculated for all patients. Estimated using Kaplan-Meier method. Log-rank tests will be used to compare among subgroups of patients.
Overall survival | Through study completion, up to 3 years
  Estimated using Kaplan-Meier method. Log-rank tests will be used to compare among subgroups of patients.

CONTACTS AND LOCATIONS:
Overall Officials: Huiying Qiu, PhD, Study Chair — The First Affiliated Hospital of Soochow University
Locations (1):
- Qiu Huiying, Suzhou, Jiangsu, China